CLINICAL TRIAL: NCT05590325
Title: Open Label, Single Arm, Two-stage Trial to Evaluate the Single and Multi-dose Pharmacokinetics and Safety of the Paediatric Dolutegravir (10 mg, Scored) Dispersible Tablet in HIV-exposed Neonates
Brief Title: Pharmacokinetics and Safety of DolutegravIr in Neonate
Acronym: PETITE-DTG
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Desmond Tutu TB Centre (Other)
Collaborators: Chiang Mai University (Other); UNITAID (Other); University of Stellenbosch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-36-SUN-MDR
Record Dates: First submitted 2022-09-06; First posted 2022-10-21 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-09

CONDITIONS: Hiv
Keywords: HIV exposed; Neonates
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: Phase I/II, open-label, single arm, two-stage pharmacokinetic and safety study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm, two-stage (Experimental): Participants will be enrolled in two stages:
  * Stage 1 will assess a single dose of the DTG-DT in two sequential cohorts: Cohort 1A (n=8) and Cohort 1B (n=8).
  * Stage 2 will assess multiple-doses of the DTG-DT and the DTG-ODF in a single cohort: Cohort 2A (n=20) DTG-DT and Cohort 2B (n=20) DTG-ODF
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — Single dose of the DTG-DT in two sequential cohorts and multiple-doses of the DTG-DT or DTG-ODF in a two cohorts.
  Qualitative Acceptability will be collected from mothers and health workers in structured discussion guides.

SUMMARY:
A Phase I/II, open-label, single arm, two-stage trial to evaluate the single and multi-dose PK and safety of DTG in HIV-exposed neonates on ARV prophylaxis. HIV-exposed term neonates born mothers with HIV on DTG-based antiretroviral therapy with a birth weight ≥2000 g who are on ARV postnatal prophylaxis will be enrolled.

DETAILED DESCRIPTION:
A Phase I/II, open-label, single arm, two-stage trial to evaluate the single and multi-dose PK and safety of DTG in HIV-exposed neonates on ARV prophylaxis. HIV-exposed term neonates born mothers with HIV on DTG-based antiretroviral therapy with a birth weight ≥2000 g who are on ARV postnatal prophylaxis will be enrolled.

Enrolment will be in two stages:

* Stage 1 will assess a single 5 mg dose of the DTG-DT in two sequential cohorts: Cohort 1A (n=8) and Cohort 1B (n=8).
* Stage 2 will assess multiple 5 mg doses of the DTG-DT and DTG-ODF in two parallel cohorts: Cohort 2A (n=20) and Cohort 2B (n=20).

Per national guidelines, all infants receive a birth HIV nucleic acid test (NAT). HIV NAT test results for the infant may or may not be available (HIV pending) at the time of study entry. HIV NAT results are typically available within 72 hours of the blood sample being taken and are checked and acted upon by the hospital HIV PMTCT service, as part of standard of care. If an HIV NAT result comes back positive whilst the neonate is on study, the neonate will not receive any further DTG doses, revert to standard of care antiretroviral therapy (ART), and be followed for safety for the duration of the study.

Primary Objectives:

* To evaluate the pharmacokinetics of dolutegravir (DTG) during the first 28 days of life in HIV-exposed term neonates (born to a mother with HIV) following administration of DTG dispersible tablet (DTG-DT) and DTG oral dispersible film (DTG-ODF)
* To determine the safety of DTG during the first 28 days of life in HIV-exposed term neonates following administration of DTG-DT and DTG-ODF

Secondary Objectives:

• To quantitatively and qualitatively assess the acceptability of DTG-DT and DTG-ODF for the neonate, the caregiver and health workers

Primary endpoints:

* DTG plasma pharmacokinetics parameters: area under the concentration time curve (AUC); maximum plasma concentration (Cmax), apparent clearance (CL/F), and trough concentration (Ctrough)
* Occurrence of the following events: adverse events of Grade 3 or higher; treatment-related adverse events of Grade 3 or higher; any adverse events

Secondary endpoints:

• Acceptability to caregivers and neonates of using DTG-DT will be measured by means of a questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Stage 1: Inclusion Criteria

  * HIV-exposed neonate (pending HIV status) born to a woman within HIV on DTG-based ART
  * Birth weight of ≥2000 g and on standard of care ARV prophylaxis

Cohort Specific Inclusion Criteria in Stage 1 must be met at Study Entry:

Cohort 1A: Infant <14 days of life Cohort 1B: Infant ≤3 days of life

Stage 2: Inclusion Criteria

* Low risk* HIV-exposed neonate (pending HIV status) born to a virologically suppressed woman on DTG-based ART

  *Neonate born to a woman with a documented plasma HIV-1 RNA result <50 copies/mL in the 4 weeks prior to delivery or between delivery and infant study entry
* Birth weight of ≥2000 g and on standard of care ARV prophylaxis

Cohort Specific Inclusion Criteria in Stage 2 must be met at Study Entry:

Cohort 2: Infant <7 days of life

Exclusion Criteria:

* • Less than 37 weeks gestational age at birth

  * Known blood group incompatibilities which can result in hemolytic disease of the newborn (e.g., Rh-negative mother, presence of antibodies on neonatal red blood cells, etc.)
  * Total bilirubin values approaching an exchange transfusion as defined by local guidelines (Section 18.2)
  * Haemoglobin value of <13.0 g/dL
  * Platelet count of less than 50,000 cells/mm3)
  * Decreased total white blood cell count (Grade 3 and above)
  * Creatinine value more than 1.3 the upper limit of normal (ULN) for gestational age and postnatal age (Grade 2 and above)
  * AST or ALT of more than 2.5 the ULN (Grade 2 and above)
  * Any other current Grade ≥3 event on the DAIDS toxicity table
  * Severe congenital abnormalities or critically ill neonates at discretion of the examining clinician
  * Receiving medicine(s) that can impact DTG pharmacokinetics (Section 8.7)
  * Participation in another clinical trial
  * HIV-infected neonates

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
In Cohort 1, PK analysis will be performed to calculate the following parameter: Cmax | first 28 days of life
  Cmax will be taken directly from the observed concentration-time data.
In Cohort 1, PK analysis will be performed to calculate the following parameter: Clast, | first 28 days of life
  Clast will be taken directly from the observed concentration-time data.
In Cohort 1, PK analysis will be performed to calculate the following parameter: Tmax | first 28 days of life
  Tmax will be taken directly from the observed concentration-time data.
In Cohort 1, PK analysis will be performed to calculate the following parameter: C24 | first 28 days of life
  C24 will be taken directly from the observed concentration-time data.
In Cohort 1, PK analysis will be performed to calculate the following parameter: AUC0-24 | first 28 days of life
  AUC0-all will be determined using the linear-up log-down trapezoidal method. Total body clearance for extravascular administration will be calculated using Dose/ AUC0-infinity. Median (range), means (standard deviations), and geometric means with 95%CI for each PK parameter will be calculated separately for Cohorts 1A and 1B, as well as for Cohort 1A/1B together.
In Cohort 1, PK analysis will be performed to calculate the following parameter: AUC0-infinity | first 28 days of life
  AUC0-infinity will be determined using the linear-up log-down trapezoidal method. Total body clearance for extravascular administration will be calculated using Dose/ AUC0-infinity. Median (range), means (standard deviations), and geometric means with 95%CI for each PK parameter will be calculated separately for Cohorts 1A and 1B, as well as for Cohort 1A/1B together.
In Cohort 1, PK analysis will be performed to calculate the following parameter: Ratio AUC0-24 / AUC0-infinity | first 28 days of life
  Ratio AUC0-24 / AUC0-infinity will be determined using the linear-up log-down trapezoidal method. Total body clearance for extravascular administration will be calculated using Dose/ AUC0-infinity. Median (range), means (standard deviations), and geometric means with 95%CI for each PK parameter will be calculated separately for Cohorts 1A and 1B, as well as for Cohort 1A/1B together.concentration-time data.
Reporting adverse events of Grade 3 or higher; treatment-related adverse events of Grade 3 or higher; any adverse events neonates following administration of DTG dispersible tablet | first 28 days of life
  Using the DAIDS toxicity table and protocol specific safety criteria
In Cohorts 2A and 2B, both non-compartmental and population PK analyses will be performed using the following parameter: Cmax | first 28 days of life
  Population means and variances of Cmax for DTG will be estimated using nonlinear mixed-effects regression models. Subject covariates will be assessed to explain sources of inter-subject PK variability.
In Cohorts 2A and 2B, both non-compartmental and population PK analyses will be performed using the following parameter: AUC0-tau | first 28 days of life
  Population means and variances of AUC0-tau for DTG will be estimated using nonlinear mixed-effects regression models. Subject covariates will be assessed to explain sources of inter-subject PK variability. Changes in DTG drug exposures in neonates following multi-doses of DTG-DT and DTG-ODF during the first 28 days of life will be estimated using the final model.
In Cohorts 2A and 2B, both non-compartmental and population PK analyses will be performed using the following parameter: CTau | first 28 days of life
  Population means and variances of CTau for DTG will be estimated using nonlinear mixed-effects regression models. Subject covariates will be assessed to explain sources of inter-subject PK variability. Changes in DTG trough concentrations in neonates following multi-doses of DTG-DT and DTG-ODF during the first 28 days of life will be estimated using the final model.
In Cohorts 2A and 2B, both non-compartmental and population PK analyses will be performed using the following parameter: Tmax | first 28 days of life
  Population means and variances of Tmax for DTG will be estimated using nonlinear mixed-effects regression models. Subject covariates will be assessed to explain sources of inter-subject PK variability.

SECONDARY OUTCOMES:
Acceptability to caregivers and neonates of using DTG-DT will be measured by means of a questionnaire | first 28 days of life
  key characteristics: Palatability, Swallowability, the device used to administer the dose, The complexity for the caregiver to prepare the dose correctly, Required dose, Need for a vehicle, Dosing frequency and duration of treatment, Selected administration devices, Primary container closure system, Actual mode of administration that reflects understanding of user instructions and feasibility of following them,
  Acceptability will be recorded by focusing on:
  Attitude of the child when presented with the formulation: facial expression, crying or smiling, reaction to drug intake, fighting drug intake, spitting out the suspension, Swallowability, i.e., ability to take the full dose, The way the caregiver prepares the dose
Qualitative acceptability data from mothers and health workers | first 28 days of life
  Data will be collected using a semi-structured discussion guide

CONTACTS AND LOCATIONS:
Overall Officials: Adrie Bekker, Prof, Principal Investigator — University of Stellenbosch
Locations (1):
- Tygerberg Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bekker A, Salvadori N, Rabie H, du Toit S, Than-In-At K, Groenewald M, Barnabas S, Ganger L, Luangcharoenkul T, Pingkarawat S, Capparelli EV, Owen A, Cressey R, Fry S, Le Roux G, Tawon Y, Kaewmalee J, Phitak T, Lallemant M, Cotton MF, Cressey TR. Safety and pharmacokinetics of dolutegravir dispersible tablets and oral films in term neonates exposed to HIV in South Africa (PETITE-DTG study): an open-label, randomised, phase 1/2 trial. Lancet HIV. 2025 Nov;12(11):e753-e762. doi: 10.1016/S2352-3018(25)00239-5. Epub 2025 Oct 8. PMID 41075812
- [Derived] Cressey TR, Salvadori N, Rabie H, du Toit S, Than-In-At K, Groenewald M, Capparelli E, Owen A, Cressey R, Lallemant M, Cotton MF, Bekker A. Single Doses of Pediatric Dolutegravir Dispersible Tablets in Neonates Support Multidosing: PETITE-Dolutegravir Study. J Acquir Immune Defic Syndr. 2025 Jun 1;99(2):195-201. doi: 10.1097/QAI.0000000000003652. PMID 39972540